CLINICAL TRIAL: NCT00504608
Title: A Multicentre, Randomised, Double-blind, Placebo-controlled Proof of Concept Study to Compare the Efficacy and Safety of r-hLIF (Emfilermin) for Improving Embryo Implantation Following in Vitro Fertilization (IVF) and Embryo Transfer (ET) in Women With Recurrent Implantation Failure
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24070
Record Dates: First submitted 2007-07-18; First posted 2007-07-20 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Infertility Implantation Failure
MeSH Terms: interventions — Leukemia Inhibitory Factor

INTERVENTIONS:
Drug: Emfilermin, recombinant human leukemia inhibitory factor (r-hLIF)

SUMMARY:
The primary objective of the study was to provide further clinical and statistical evidence of the efficacy of r-hLIF, in comparison with placebo, administered during the luteal phase after IVF and ET for improving embryo implantation in infertile women with a history of at least 2 implantation failures following transfer of fresh embryos. The secondary objective of the study was to assess the safety profile of r-hLIF in the proposed indication.

ELIGIBILITY:
Inclusion Criteria:

1. Pre-menopausal woman aged 21-37 years inclusive at time of consent.
2. Infertile woman justifying IVF-ET treatment and wishing to conceive.
3. The presence of both ovaries.
4. Current body mass index (BMI) of ≥ 20 & ≤ 30 kg/m2
5. Early follicular phase (cycle day 2-5) serum FSH levels ≤ 10 IU/L. If two determinations are available, at least one should be < 10 IU/L.
6. History of:

   * ≥ 2 ART cycles with adequate stimulation that led to the transfer of at least two or more fresh Grade A or B embryos, but did not result in implantation or
   * ≥ 3ART cycles with adequate stimulation that led to the transfer of at least one fresh Grade A or B embryo from a cohort with one additional Grade A or B embryo, but did not result in implantation
7. Normal male partner's semen analysis according to standard WHO criteria. Male partner's semen analysis must be suitable for IVF (ICSI not allowed). Donor sperm is allowed.
8. Normal cervical cytology within 3 years prior to starting GnRH-agonist therapy.
9. At least one wash-out cycle (defined as ≥ 30 days since the last dose of clomiphene citrate or gonadotrophin treatment) since the last ART cycle and/or clomiphene citrate or gonadotrophin treatment, prior to starting GnRH-agonist therapy.
10. Negative pregnancy test within 7 days prior to starting GnRH-agonist therapy.
11. Willingness and ability to comply with the protocol for the duration of the study.
12. Written informed consent given prior to any study-related procedure not part of the patient's normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.

Exclusion Criteria:

1. Known to be positive for Human Immunodeficiency Virus, Hepatitis B or C Virus.
2. History of any liver disease.
3. Any one of the following parameters above the upper limit of normal at the prestudy visit: AST, ALT, Alkaline phosphatases, gamma GT, alpha GST, bilirubin.
4. Any clinically significant systemic disease.
5. Any significant allergic disease.
6. Presence of an uncontrolled clinically significant medical condition including infection) as determined by the investigator.
7. History of ART biochemical pregnancy.
8. Any cause of infertility that would justify ICSI treatment
9. Presence of another known cause of previous ART failure other than recurrent implantation failure.
10. Uterine cavity with abnormalities which, in the investigator's opinion, could impair embryo implantation or pregnancy outcome, as assessed by US examination performed within 6 months prior to starting GnRH-agonist therapy.
11. More than one previous failed ART cycle, where "failed" is defined as cancellation of administration of hCG or poor response to gonadotrophin stimulation (defined as retrieval of 3 oocytes or less).
12. Any history of difficulties in ET procedure (i.e. requiring general anaesthetic e.g. due to position of cervix).
13. Abnormal undiagnosed gynaecological bleeding.
14. Any contraindication to being pregnant and/or carrying pregnancy to term.
15. Presence of any medical condition for which the use of gonadotrophin preparations or progesterone is contra-indicated.
16. Known allergy to Escherichia coli derived pharmaceutical products.
17. Known allergy or hypersensitivity to gonadotrophin preparations.
18. Known intolerance or allergy to paracetamol (acetaminophen).
19. Active substance abuse.
20. Previous LIF therapy in the same indication.

Ages: 21 Years to 37 Years | Sex: Female
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2003-04; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Improvement of embryo implantation and safety | Various

SECONDARY OUTCOMES:
Implantation rate, all pregnancy rateand number of live births. | Various

CONTACTS AND LOCATIONS:
Overall Officials: Paul Barrière, M.D., Principal Investigator — Bourn Hall Clinic, Bourn Hall, High Street, Bourn, Cambridge CB3 7TR